CLINICAL TRIAL: NCT02306135
Title: Identifying Mechanisms of Resistance to mTOR Inhibitors in Cancer
Status: Terminated | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: D15036
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
Keywords: Cancer; Tumor; Everolimus; mTOR; Temsirolimus; Sirolimus; Rapamycin
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Tumor biopsy and surgical specimens obtained through routine clinical procedures and archived in the institution's Pathology tissue bank will be used for DNA extraction for genetic analysis.
  Blood samples collected prospectively will be used to extract plasma and leukocytes, which will be used to extract DNA for genetic analysis.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: n/a- this is an observational study

SUMMARY:
mTOR kinase is part of the mTORC1 complex that promotes cap-dependent protein translation, and part of the mTORC2 complex that activates AKT. Everolimus (Afinitor) is an allosteric inhibitor of mTOR that suppresses mTORC1 activity. Everolimus is FDA-approved for the treatment of ER+/HER2- breast cancer (in combination with exemestane), renal cell carcinoma, subependymal giant cell astrocytoma (SEGA), and neuroendocrine tumors of pancreatic origin (PNET), and is currently being tested in ongoing clinical studies in other indications. While everolimus-based therapies elicit anti-cancer effects, most cancers ultimately progress and exhibit everolimus resistance. This study will evaluate genetic mechanisms of resistance to everolimus.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment with everolimus (as a single-agent or in combination) for any malignancy for ≥3 months.
2. A- Patients who are scheduled to undergo a clinically indicated tumor biopsy (as standard of care, or as part of another study) within 5 years following cancer progression on everolimus are eligible.

   B- Patients who already had such a biopsy procedure performed are eligible. Tumors biopsied shortly after progression on everolimus are strongly preferred.
3. Excess tumor tissue from biopsy must be available for molecular analysis. This will include tumor tissue sufficient to make ≥5 five-micron sections; more tumor tissue is preferred.
4. Patients currently seen at Dartmouth-Hitchcock Medical Center must be capable and willing to provide informed written consent for study participation. Patients who are no longer seen at DHMC will not be consented for use of archived tissues and data.
5. For patients currently seen at Dartmouth-Hitchcock Medical Center, patients must be willing to provide an extra 10-20 mL of blood during a routine, clinically indicated blood draw procedure.

Exclusion Criteria:

none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with everolimus for any cancer type.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Mutations in genes encoding components of the mTOR pathway that are detected in post-everolimus tumors but not pre-everolimus tumors. | 1 year

SECONDARY OUTCOMES:
Mutations detected in plasma DNA that are present in the post-everolimus tumor but not the pre-everolimus tumor. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Todd W Miller, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States